CLINICAL TRIAL: NCT01548898
Title: The Efficacy of Laser Assisted Hair Removal in the Treatment of Acne Keloidalis Nuchae; a Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Abdel hay, lecturer of Dermatology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nd-YAG laser in AKN
Record Dates: First submitted 2012-02-29; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Acne Keloidalis Nuchae
MeSH Terms: conditions — Acne Keloid | interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Nd-YAG laser — All patients received 5 sessions (4 weeks apart) of long pulsed nd-YAG laser assisted hair removal on the affected area, emitting 1064 nm, with a fluence of 35-45 J/cm2 and pulse duration 10-30 msec adjusted to skin type and hair thickness. Laser was applied to all papules and plaques.

SUMMARY:
Laser causes elimination and miniaturization of hair shafts that are the principal contributor to inflammation in Acne Keloidalis Nuchae (AKN).

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from AKN

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Global response to treatment | 6 months

SECONDARY OUTCOMES:
Patient satisfaction | 6 months